CLINICAL TRIAL: NCT04329299
Title: Use of Blood Biomarkers to Predict Gastric Cancer Risk
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other); MiRXES Pte Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 2012/00737
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-03

CONDITIONS: Stomach Neoplasm
Keywords: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 15 ml of Blood sample collected from each study participant, will be processed to extract serum, plasma and white blood cells.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Biomarkers Analyses: 15 ml of blood sample will be obtained from each study participant, for blood-based biomarkers analyses.
  Interventions: Diagnostic Test: blood-based biomarkers analyses

INTERVENTIONS:
Diagnostic Test: blood-based biomarkers analyses — Analyses of H. pylori antibodies/pepsinogen levels, micro RNAs (miRNAs) or blood-based protein markers levels in participants' blood samples

SUMMARY:
This study aims to develop a cost-effective screening strategy for the Singapore population by targeted screening of people who have a high risk of stomach cancer, in order to detect early signs of the disease at a stage that can be prevented or cured. Often, patients only consult their doctors when they have advanced symptoms, by which time the cancer may be at a difficult to treat, or incurable stage.

Using costs in the Singapore health system as well as local population risk profiles and demographics, our previous study demonstrated that screening of high-risk groups is cost-effective and a panel of serum makers was effective in differentiating high-risk from low-risk individuals. This study aims to validate the predictive value of various blood biomarkers, such as that of antibodies against Helicobacter pylori, pepsinogen levels, micro RNAs (miRNAs) and blood-based protein markers in participants who have been scheduled to undergo upper gastrointestinal (GI) endoscopy for clinical reasons. If successful, the marker can be used to stratify population into different risk groups and various screening systems can be provided according to different risk level. This will reduce the number of annual invasive screening examinations required to detect early gastric cancer (GC), thereby rendering it cost-effective to generalize as clinical practice in Singapore.

DETAILED DESCRIPTION:
Objectives:

This study aims to

1. Validate the predictive value of various blood biomarkers, including the panel of antibodies against H.pylori and pepsinogen levels, micro RNAs (miRNAs) and blood-based protein markers in a prospective cohort study involving 8000 participants who have been referred for upper for predicting gastric cancer risk.
2. Record the number of participants who are diagnosed with gastric cancer, including high grade dysplasia, carcinoma in-situ and adenocarcinoma.
3. Develop a cost-effective screening strategy based on 1 and 2.

Study Design This is a prospective cohort study involving 8000 subjects who are referred for upper GI endoscopy for standard clinical indications. Blood will be drawn from subjects for blood tests, including antibodies against H. pylori, pepsinogen levels, specific miRNA levels, blood-based protein markers, before undergoing an upper GI endoscopy for clinical reasons. Subjects will be monitored for a period of 10 years via verification with the National Registry of Diseases Office (NRDO) of Singapore. The correlation between the blood test results and findings from the clinical endoscopy or NRDO database verification will be analyzed to determine the predictive value.

Enrolment Patients undergoing upper gastrointestinal endoscopy will be considered for enrolment provided they meet the inclusion and exclusion criteria. 8000 subjects will be enrolled. The Patient Informed Consent Form will be discussed with the patient. If acceptable, the form will be signed by the patient, Principal Investigator and witness if applicable. The subject will be assigned initials and a number in the order in which they were enrolled. Subjects will also be asked to provide information on demographics, family history of gastric cancer, diet, medical history, and lifestyle habits. The data will be captured in a comprehensive database.

Blood Collection 15 mls of blood will be drawn from each subject. Serum, plasma and white blood cells will be extracted.

Analyses

1. Sera will be assayed for antibodies against H. pylori, Pepsinogen I and II levels to derive H. pylori status and pepsinogen index. Participants will be classified into 4 groups, A, B, C and D, according to H. pylori status and pepsinogen Index. Group A includes subjects negative for both H. pylori antibodies and pepsinogen atrophic gastritis (PGA). Group B subjects will be negative for PGA and positive for H.pylori antibodies. Group C subjects will be positive for both tests. Finally, Group D subjects will be positive for PGA and negative for H. pylori antibodies. The incidence rate and relative risk of gastric cancer as determined by the findings of subjects' clinical gastroscopies or verification with NRDO will be calculated.
2. Total RNA from serum or plasma will be isolated and the expression levels of miRNAs will be determined. The final miRNA expression levels after normalization of both technical and biological variations are analyzed with multiple statistical methods to identify panels of miRNAs with the highest discriminatory power between healthy and disease states. Each participant will be assigned a score based on miRNA expression profile, indicating the possibility of having GC. The result will be compared with endoscope and histology result which is the gold standard for diagnosis of GC. We will compare the performance of our miRNA panel with other serum markers including H. pylori status and pepsinogen levels.
3. Levels of 10 blood-based protein markers (determined from systematic review) will be analyzed from sera through ELISAs (enzyme-linked immunosorbent assay). Subsequent statistical multivariate analysis may be applied to generate a biomarker panel with a superior diagnostic performance compared to the conventional blood-based biomarkers for gastric cancer.

Sample Size Calculation In our previous case-control study, 10% of the control group had pepsinogen (PG) determined atrophic gastritis, and the odds ratio (95%CI) for the risk of developing gastric cancer was 4.02 (2.56-6.30) compared with subjects who had no PG atrophic gastritis. A minimum of 47 gastric cancer cases are required to evaluate the PG-H. Pylori panel in the prediction of gastric cancer risk (with odds ratio 3.5) at power of 90% and p-value <0.05. Based on the estimated gastric cancer prevalence rate among NUH patients of the gastroenterology and upper GI surgery clinics of 0.6%, a cohort size of 8000 subjects will be needed.

Statistical Analysis The chi-square test and the t-test will be used to compare the distributions of selected demographic, lifestyle and other risk factors between cases and controls. The logistic regression method will be used to examine the associations between blood markers measured and risk of gastric cancer. Statistical computing will be carried out using the SPSS 19. The statistical significance level is set at two-sided P value of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is greater than 40 years of age.
2. The subject is scheduled to undergo an endoscopy because of medical indication.
3. The subject must have personally signed and dated the patient informed consent form indicating that he/she has been informed of all pertinent aspects of the study.
4. The subject must be willing and able to comply with all study procedures.

Exclusion Criteria:

1. The subject who is unable to undergo gastroscopy.
2. The subject with previous total or partial gastrectomy.
3. The subject has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may interfere with the interpretation of study results and in the judgment of the investigator would make the subject unsuitable for entry into the study.
4. The subject is unwilling or unable to provide signed informed consent.
5. The subject who is pregnant.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to the participating study sites for upper GI endoscopy for standard clinical indications.
Sampling Method: Non-Probability Sample
Enrollment: 6862 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2016-05-29 (Actual); Study Completion 2016-05-29 (Actual)

PRIMARY OUTCOMES:
Gastric cancer | 10 years
  Number of patients who develop gastric cancer, including high grade dysplasia, carcinoma in-situ and adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Jianyi Koh, MBBS, MMed, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore, Singapore

REFERENCES:
- [Background] Dan YY, So JB, Yeoh KG. Endoscopic screening for gastric cancer. Clin Gastroenterol Hepatol. 2006 Jun;4(6):709-16. doi: 10.1016/j.cgh.2006.03.025. PMID 16765306
- [Background] Miki K. Gastric cancer screening by combined assay for serum anti-Helicobacter pylori IgG antibody and serum pepsinogen levels - "ABC method". Proc Jpn Acad Ser B Phys Biol Sci. 2011;87(7):405-14. doi: 10.2183/pjab.87.405. PMID 21785258
- [Background] Cortez MA, Bueso-Ramos C, Ferdin J, Lopez-Berestein G, Sood AK, Calin GA. MicroRNAs in body fluids--the mix of hormones and biomarkers. Nat Rev Clin Oncol. 2011 Jun 7;8(8):467-77. doi: 10.1038/nrclinonc.2011.76. PMID 21647195
- [Background] Song JH, Meltzer SJ. MicroRNAs in pathogenesis, diagnosis, and treatment of gastroesophageal cancers. Gastroenterology. 2012 Jul;143(1):35-47.e2. doi: 10.1053/j.gastro.2012.05.003. Epub 2012 May 10. PMID 22580099
- [Derived] So JBY, Kapoor R, Zhu F, Koh C, Zhou L, Zou R, Tang YC, Goo PCK, Rha SY, Chung HC, Yoong J, Yap CT, Rao J, Chia CK, Tsao S, Shabbir A, Lee J, Lam KP, Hartman M, Yong WP, Too HP, Yeoh KG. Development and validation of a serum microRNA biomarker panel for detecting gastric cancer in a high-risk population. Gut. 2021 May;70(5):829-837. doi: 10.1136/gutjnl-2020-322065. Epub 2020 Oct 7. PMID 33028667
- [Derived] Bibault JE, Chang DT, Xing L. Development and validation of a model to predict survival in colorectal cancer using a gradient-boosted machine. Gut. 2021 May;70(5):884-889. doi: 10.1136/gutjnl-2020-321799. Epub 2020 Sep 4. PMID 32887732